CLINICAL TRIAL: NCT05087615
Title: Effects of Ondansetron, Metoclopramide and Granisetron on Perioperative Nausea and Vomiting in Patients Undergone Bariatric Surgery: a Randomized Clinical Trial
Brief Title: Effects of Ondansetron, Metoclopramide and Granisetron on Perioperative Nausea and Vomiting in Patients Undergone Bariatric Surgery
Acronym: PONV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Manoochehr Ebrahimian, Principal Investigator, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ManoochehrEbrahimian
Record Dates: First submitted 2021-10-08; First posted 2021-10-21 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Bariatric Surgery Candidate; Perioperative Complication; Nausea; Vomiting, Postoperative; Drug Effect
Keywords: Bariatric Surgery; Post-operative nausea or vomiting; Sleeve Gastrectomy; Ondansetron; Metoclopramide; Granisetron
MeSH Terms: conditions — Nausea; Postoperative Nausea and Vomiting; Vomiting | interventions — Metoclopramide; Ondansetron; Granisetron

STUDY DESIGN:
Intervention Model Description: the patients were divided into five parallel groups including control and study groups.
  Group 1: Patients who did not receive any antiemetic during hospitalization (NA).
  Group 2: Patients receiving metoclopramide alone (MA). Group 3: Patients who received ondansetron only. (OA) Group 4: Patients receiving a combination of metoclopramide and ondansetron (MO).
  Group 5: Patients who received granisetron alone (GA).
Who Masked: Participant, Care Provider, Investigator
Masking Description: After taking informed consent, patients enrolled in the groups. Each group had 26 members, and the subjects were unaware of which group they had been assigned. Also, the investigators weren't aware of the treatment assignment until the end of the trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Control (No Intervention): Patients who did not receive any antiemetic during hospitalization (NA).
- MA (Experimental): Patients receiving metoclopramide alone (MA).
  Interventions: Drug: Metoclopramide
- OA (Experimental): Patients who received ondansetron only (OA).
  Interventions: Drug: Ondansetron
- MO (Experimental): Patients receiving a combination of metoclopramide and ondansetron (MO).
  Interventions: Drug: Metoclopramide and Ondanteron
- GA (Experimental): Patients who received granisetron alone (GA).
  Interventions: Drug: Granisetron

INTERVENTIONS:
Drug: Metoclopramide — This groups only received metoclopramide 0.2 mg/kg IV Bid as antiemetic in the postoperative period.
  Other Names: Plasil
  Arms: MA
Drug: Ondansetron — This groups only received ondansetron 8 mg IV Bid as antiemetic in the postoperative period.
  Arms: OA
Drug: Metoclopramide and Ondanteron — This groups received both metoclopramide 0.2 mg IV Bid and ondansetron 8 mg IV/Bid as antiemetics in the postoperative period.
  Arms: MO
Drug: Granisetron — This groups only received granisetron 2 mg IV Bid as antiemetic in the postoperative period.
  Arms: GA

SUMMARY:
Post-operative nausea and vomiting (PONV) is one of the leading causes of patient morbidity after laparoscopic bariatric surgeries. A wide variety of complications related to PONV has been described, such as prolonged length of stay (LOS) in hospital, unnecessary readmissions, delay in oral intake, and bad experience for patients. Although several antiemetic regimens have been tried so far in different studies, the incidence of PONV is not significantly lowered, and it seems that it is impossible to totally eliminate it. On the other hand, the implementation of Enhanced Recovery After Surgery (ERAS) has greatly reduced the incidence of PONV and LOS. Therefore, a combination of ERAS and multiple antiemetic regimens is currently used to reduce the incidence of PONV. Nevertheless, the optimal regimen has not been found yet, and many trials are conducting to find out the best antiemetic regimen. In this randomized clinical trial, we compare four different combined and single regimens alongside the implementation of ERAS to show which regimen is more effective.

DETAILED DESCRIPTION:
After being approved by Iran National Committee for Ethics in Biomedical Research (IR.SBMU.MSP.REC.1399.784), a randomized clinical controlled trial was started with 130 patients in five groups. All the patients were proper candidates for laparoscopic bariatric surgeries, and structured informed consent was obtained from all participants.

All the operations were performed by board certified advanced laparoscopic surgeons in a minimally invasive educational center. All bariatric surgery was performed in our standardized institutional protocols as well as preoperative and postoperative care. Sleeve Gastrectomy (SG) surgeries were performed by using 44Fr Tubes.

To calculate the sample size in the clinical trial, we used the ANCOVA method with web-based tools. Twenty-six patients were estimated for each group. Patients were divided into five groups:

Group 1: Patients who did not receive any antiemetic during hospitalization (NA).

Group 2: Patients receiving metoclopramide alone (MA). Group 3: Patients who received ondansetron only. (OA) Group 4: Patients receiving a combination of metoclopramide and ondansetron (MO).

Group 5: Patients who received granisetron alone (GA). All patients were undergone ERAS protocols. In cases where the patient had PONV (including Group 1), intravenous Metoclopramide 0.2mg (Stat and BiD) was used as a rescue antiemetic.

To reduce the incidence of bias and confounding factors, all anesthetics and antiemetics used were provided from the same brand for each drug (see Appendix).

Patients with severe or moderate gastritis or duodenitis on esophagogastroduodenoscopy were excluded from the study, but patients with mild gastritis or positive rapid urease test on endoscopy, were treated for two weeks with three drugs of pentazole, amoxicillin, and metronidazole, and if the respiratory urease test was negative, they were included in the study and in refractory cases of H. Pylori, they were excluded. According to the American Society of Anesthesiologists (ASA) classification, patients with severe respiratory or cardiovascular problems (ASA III or higher) or a history of gastric or small bowel surgery were also excluded. Patients who underwent simultaneous cholecystectomy with bariatric surgery were also excluded.

ELIGIBILITY:
Inclusion Criteria:

* BMI>40
* Only bariatric operations
* mild or moderate surgical risk
* without any previous gastrointestinal problems
* no previous gastrointestinal surgery

Exclusion Criteria:

* Moderate or severe gastritis or duodenitis
* GERD
* lack of H. Pylori eradication
* concurrent cholecystectomy
* Dissatisfaction during study

Ages: 13 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-08-21 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
Change PONV | PONV has been measured in day one, and two of admission
  reduction in the incidence of postoperative nausea/vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Loghman Hakim Hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
All the data and analytic works will be available for interested persons.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: from February 2022
Access Criteria: Everyone with verified institutional email.

REFERENCES:
- [Background] Naeem Z, Chen IL, Pryor AD, Docimo S, Gan TJ, Spaniolas K. Antiemetic Prophylaxis and Anesthetic Approaches to Reduce Postoperative Nausea and Vomiting in Bariatric Surgery Patients: a Systematic Review. Obes Surg. 2020 Aug;30(8):3188-3200. doi: 10.1007/s11695-020-04683-1. PMID 32415635
- [Background] Therneau IW, Martin EE, Sprung J, Kellogg TA, Schroeder DR, Weingarten TN. The Role of Aprepitant in Prevention of Postoperative Nausea and Vomiting After Bariatric Surgery. Obes Surg. 2018 Jan;28(1):37-43. doi: 10.1007/s11695-017-2797-0. PMID 28674839
- [Background] Fathy M, Abdel-Razik MA, Elshobaky A, Emile SH, El-Rahmawy G, Farid A, Elbanna HG. Impact of Pyloric Injection of Magnesium Sulfate-Lidocaine Mixture on Postoperative Nausea and Vomiting After Laparoscopic Sleeve Gastrectomy: a Randomized-Controlled Trial. Obes Surg. 2019 May;29(5):1614-1623. doi: 10.1007/s11695-019-03762-2. PMID 30734195
- [Background] Moussa AA, Oregan PJ. Prevention of postoperative nausea and vomiting in patients undergoing laparoscopic bariatric surgery--granisetron alone vs granisetron combined with dexamethasone/droperidol. Middle East J Anaesthesiol. 2007 Jun;19(2):357-67. PMID 17684876